CLINICAL TRIAL: NCT07045766
Title: FaibaLite - Reduce Weight, One Bite at a Time
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: DCB Research AG (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FaibaLite
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Nutritional and Metabolic Diseases
Keywords: Chewing gum; Galactooligosaccharides; GOS (Galactooligosaccharides); Intestinal microbiome; Gut microbiota
MeSH Terms: conditions — Nutritional and Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Mono-centre, single-arm, open-label feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FibreGum Intervention Group (Experimental): Participants chew one fiber-containing gum (FibreGum) three times daily (morning, noon, and evening) for at least 20 minutes each, over two months, with the option to extend the intervention to three months.
  Interventions: Dietary Supplement: FibreGum chewing gum

INTERVENTIONS:
Dietary Supplement: FibreGum chewing gum — Chewing gum containing galactooligosaccharides (GOS), delivering a total daily dose of 3 g of dietary fiber.

SUMMARY:
This study aims to evaluate the suitability of a fiber-enriched chewing gum as a practical and accessible approach to support healthy body weight management.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Healthy adults aged 18 to 65 years (inclusive), as determined by the investigator
* BMI of 23 to 40 kg/m2 (inclusive)
* Living in Switzerland
* Ability and willingness to follow the study protocol (e.g., cognitive capacity for compliance, gum chewing)
* Access and willingness to use an electronic device (e.g., mobile phone, computer or tablet)
* Access to a scale to self-report weight

Exclusion Criteria:

* Current weight loss therapy with Glucagon-like Peptide 1 (GLP-1) agonists or other non-prescription products (at investigator's discretion)
* Treatment with a GLP-1 agonist within the past 2 months
* Initiation/Discontinuation of nicotine product use (>1 nicotine product per day, e.g., (e-)cigarette, gum) within the last 2 months (at investigator's discretion)
* Significant change in medication within the last 2 months (at investigator's discretion)
* Unable to chew gum 3 times daily (e.g. due to dental issues, at investigator's discretion)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Composite primary endpoint: Feasibility of conducting the study based on participant adherence rate, user acceptance score, and dropout rate | Up to 3 months (end of chewing phase)
  Feasibility will be assessed as a composite endpoint including the following parameters among healthy adults:
  * Participant adherence rate (percentage of recommended chewing performed)
  * User acceptance score (based on questionnaire)
  * Dropout rate (percentage of participants who discontinue the study prematurely)

SECONDARY OUTCOMES:
Duration of intervention | Up to 3 months after study start
  Duration of the study intervention, e.g. the willingness to continue FibreGum consumption for an additional month after 2 months of intervention
Reduction in body weight (%) | 2 or 3 months
  Reduction in percent of body weight between baseline and end of intervention
Change in body composition (body fat) | 2 or 3 months
  Difference in body fat* (if available) between baseline and end of intervention
  *This read-out is voluntary for participants willing to come to the investigational site according to Table of Assessment
Change in body composition (lean mass) | 2 or 3 months
  Difference in lean mass* (if available) between baseline and end of intervention
  *This read-out is voluntary for participants willing to come to the investigational site according to Table of Assessment
Change in body composition (muscle mass) | 2 or 3 months
  Difference in muscle mass* (if available) between baseline and end of intervention
  *This read-out is voluntary for participants willing to come to the investigational site according to Table of Assessment
Change in gut microbiota alpha-diversity | 2 months
  Change in microbial community diversity (alpha diversity) from baseline to timepoint 2, assessed by established diversity metrics
Change in gut microbiota beta-diversity | 2 months
  Change in microbial community composition from baseline to timepoint 2, assessed by beta diversity metrics
Change in differential abundance of gut microbiota | 2 months
  Change in the relative abundance of specific bacterial taxa between baseline and timepoint 2, assessed by metagenomic sequencing
Changes in body weight during follow-up | 1 or 2 months
  Changes in body weight from completion of intervention to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Balmer, Prof. med., Principal Investigator — Department of Biomedical Research, University of Bern
Locations (1):
- Department of Biomedical Research, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No